CLINICAL TRIAL: NCT05316779
Title: Perioperative Cardiac Arrest: an Observational Mono-centre 8-year Assessment of Outcome
Brief Title: Perioperative Cardiac Arrest and Outcome
Acronym: POCA
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02330
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Heart Arrest; Anesthesia
Keywords: Cardiac arrest; Perioperative cardiac arrest; Neurological outcome; Quality of Life; In-hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With ethical approvement, the investigators want to assess the incidence, circumstances and outcomes of patients with perioperative cardiac arrests over a period of 8 years.

Currently, there is little data and information about a cardiovascular arrests during anesthesia. Little is also known about the health-related quality of life afterwards. In the investigators research project, the investigators want to find out if there are, for example, specific factors that cause cardiovascular arrests and factors that can improve the chances of survival after a cardiovascular arrest. The investigators are also looking for possible factors and measurements that can minimize or even prevent future events during anesthesia.

DETAILED DESCRIPTION:
A perioperative cardiac arrest is a special form of in-hospital cardiac arrest. It was claimed that perioperative cardiac arrests are under-investigated. The spare existing data suggest incidences of perioperative cardiac arrest to be between 0.5 - 3 per 10.000 for adult patients and 2 - 10 per 10.000 for paediatric patients. Data on circumstances, predictors and outcomes of perioperative cardiac arrest are rare, especially for paediatric patients. Some reports suggest that incidence is negatively associated with a country's higher development. As no Swiss data is available on this topic, this retrospective audit aims to bridge the knowledge gap and finally intends to make clinicians aware of potential risks or contributing factors of survival, which might raise safety for all patients undergoing procedures under anaesthesia.

The investigators will include all patients of all ages with a perioperative cardiac arrest at Bern University Hospital from 1st January 2015 until 31st December 2021 (7 year observational period).

ELIGIBILITY:
Inclusion Criteria is a perioperative cardiac arrest between 1st January 2015 and 31st December 2021 at Bern University Hospital.

A perioperative cardiac arrest is defined as:

* ≥5 chest compressions (direct, mechanical or extracorporeal Cardiopulmonary Resuscitation (CPR))
* and/or defibrillation (unsynchronised direct current (DC) shock for ventricular fibrillation (VF) or pulseless ventricular tachycardia (pVT) either - external or internal defibrillation with manual or Automated External Defibrillation (AED), shocks by implanted cardioverter defibrillators (ICDs) for VF/pVT, precordial thump)
* In a patient having a procedure under the care of an anaesthesia team (nurse or anaesthesiologist) at the Bern University Hospital: General anaesthesia, regional anaesthesia/ analgesia, sedation, local anaesthesia or monitored anaesthesia care
* Regional block performed by anaesthesiologist outside of operating room
* Obstetric analgesia including remifentanil patient-controlled analgesia (PCA).

Exclusion Criteria:

* A perioperative cardiac arrest before 1st January 2015 or after 31st December 2021
* <5 chest compressions (direct, mechanical or extracorporeal Cardiopulmonary Resuscitation (CPR))
* All in-hospital cardiac arrests, that occur without being under anaesthesia care
* Patients already admitted to a hospital with a cardiac arrest (out-of hospital cardiac arrests)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will include all patients of all ages with a perioperative cardiac arrest at Bern University Hospital from 1st January 2015 until 31st December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) | 60 minutes
  Number of patients with a Return of spontaneous circulation (ROSC) during resuscitation

SECONDARY OUTCOMES:
Sustained ROSC | 60 minutes
  Number of patients with a Return of spontaneous circulation during resuscitation over 20 minutes
Survival post-anaesthesia care unit or intensive care unit | 24 hours
  Number of patients with a Survival to post-anaesthesia care unit (PACU) or intensive care unit (ICU)
Survival to hospital discharge | 4 weeks
  Number of patients with a Survival to hospital discharge
SF-12 after hospital discharge | 1 month
  Health-related quality of life according (HRQOL) the Short Form Survey (SF-12) after hospital discharge
CPC after hospital discharge | 1 month
  Neurological status according Clinical Performance Category (CPC) after hospital discharge
SF-12 3 month after cardiac arrest | 3 months
  Health-related quality of life (HRQOL) according the Short Form Survey (SF-12) at 3 months after the peri-operative cardiac arrest
CPC 3 month after cardiac arrest | 3 months
  Neurological status according Clinical Performance Category (CPC) at 3 months after the peri-operative cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Prof, Study Director — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No